CLINICAL TRIAL: NCT07113834
Title: Characteristics of Ankylosing Spondylitis Associated Uveitis: A Retrospective Study in Egyptian Patients
Brief Title: Characteristics of Ankylosing Spondylitis Associated Uveitis
Acronym: uveitis
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Elsayed Mohamed Saad, Lecturer, Benha University
Other Study IDs: Ankylosing
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2023-09

CONDITIONS: Uveitis
Keywords: Ankylosing Spondylitis; Uveitis
MeSH Terms: conditions — Uveitis; Spondylitis, Ankylosing | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Adalimumab — A tumor necrosis factor-alpha (TNF-α) inhibitor used as a biologic agent for the treatment of ankylosing spondylitis. Administered subcutaneously as part of systemic immunomodulatory therapy.
Drug: Systemic corticosteroids — Oral or intravenous corticosteroids (e.g., prednisolone) used to suppress systemic inflammation in cases of active AS or severe uveitis.

SUMMARY:
This study aims to understand the clinical characteristics associated with AAU in Egyptian AS patients, and the prognostic factors, in terms of the Corrected Distance Visual Acuity (CDVA).

DETAILED DESCRIPTION:
This is a one-year retrospective cohort study conducted at the Spine and Ophthalmology Clinics of Benha University - Faculty of Medicine, Egypt, between September 2023 and August 2024. The study aims to characterize the clinical features and identify prognostic factors affecting visual outcomes in patients with Ankylosing Spondylitis-associated Anterior Uveitis (ASAAU).

Patients included in this study were Egyptian nationals who initially presented to the Spine Clinic with systemic symptoms of ankylosing spondylitis (AS) and were subsequently referred to the Ophthalmology Clinic due to ophthalmic complaints. Only patients who were confirmed to have both AS (diagnosed according to the Modified New York criteria and radiographic imaging) and anterior uveitis (confirmed by slit-lamp examination and supported by Optical Coherence Tomography [OCT] and Fluorescein Angiography [FA]) were enrolled.

The final sample included 26 eyes from 22 patients who fulfilled the inclusion criteria. Patients were excluded if they were non-Egyptian, had other systemic autoimmune or immunologic conditions, had uveitis due to secondary causes, had undergone ocular surgeries, did not receive uveitis treatment, were lost to follow-up, or had incomplete medical records.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian nationality.

Age: ≥ 18 years.

Confirmed diagnosis of Ankylosing Spondylitis (AS) according to the Modified New York Criteria, including:

Clinical symptoms (e.g., chronic inflammatory back pain, reduced lumbar motion, reduced chest expansion)

Radiographic evidence of sacroiliitis.

Confirmed diagnosis of Acute Anterior Uveitis (AAU) based on:

Ophthalmologic examination (e.g., slit-lamp biomicroscopy)

Ancillary testing (e.g., Optical Coherence Tomography [OCT] and/or Fluorescein Angiography [FA]).

Presentation to the Spine Clinic of Benha University - Faculty of Medicine between September 2023 and August 2024 with ophthalmic complaints, subsequently referred to the Ophthalmology Clinic.

Complete medical and ophthalmologic records available.

Received treatment for both AS and AAU.

At least one follow-up visit after initiation of treatment.

Exclusion Criteria:

* Non-Egyptian patients.

History of other systemic autoimmune or immunological diseases (e.g., sarcoidosis, Behçet's disease, systemic lupus erythematosus).

Uveitis due to non-autoimmune secondary causes (e.g., infectious uveitis, trauma-related uveitis).

History of ocular surgery prior to the episode of AAU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study included a retrospective cohort of 22 Egyptian patients (26 eyes) diagnosed with Ankylosing Spondylitis-associated Acute Anterior Uveitis (ASAAU), who were referred to the Ophthalmology Clinics of Benha University - Faculty of Medicine from the Spine Clinic at the same institution between September 2023 and August 2024. The cohort was composed of adult patients who met the Modified New York Criteria for AS and had documented ophthalmic symptoms confirmed as AAU through clinical and imaging evaluation. All included patients had complete follow-up data and received appropriate treatment for both AS and uveitis.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Corrected Distance Visual Acuity (CDVA) | Baseline and 3-month follow-up
  CDVA was assessed at baseline (initial presentation) and after treatment (follow-up average of 3 months), using the Logarithm of the Minimum Angle of Resolution (logMAR) scale. Improvement or deterioration in CDVA was evaluated in relation to clinical characteristics, treatment modalities, and complication development.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, Cairo Governorate, Egypt